CLINICAL TRIAL: NCT02293226
Title: Comparison of Four Video-laryngoscopes During Pediatric Intubation During Simulated Resuscitation
Brief Title: Video-laryngoscopy During Chest Compression
Acronym: VIDEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/19
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest; Intubation, Endotracheal
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child ETI with chest compressions (Experimental): endotracheal intubation (ETI) during child mannikin resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: CoopDech; Device: CoPilot; Device: Intubrite; Device: Vividtrack
- Infant ETI with chest compressions (Experimental): endotracheal intubation (ETI) during infant mannikin resuscitation with uninterrupted chest compressions
  Interventions: Device: CoopDech; Device: CoPilot; Device: Intubrite; Device: Vividtrack

INTERVENTIONS:
Device: CoopDech — Video-laryngoscopy 1
  Other Names: Coopdech Video Laryngoscope Portable VLP-100
Device: CoPilot — video-laryngoscopy 2
  Other Names: CoPilot VideoLaryngoscope
Device: Intubrite — Video-laryngoscopy 3
  Other Names: Intubrite Video Laryngoscope System VLS 6600
Device: Vividtrack — video-laryngoscopy 4

SUMMARY:
The investigators will compare the success rates and time to successful intubation of endotracheal intubation during simulated pediatric and infant resuscitation with and without chest compression using four different video-laryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* Minimum 1 year of work experience in nursing

Exclusion Criteria:

* Not meet the above criteria
* Wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | 1 day
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
Cormack-Lehan scale | 1 day
  self reported Cormack-Lehan scale during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland